CLINICAL TRIAL: NCT01645046
Title: The Effects of Coenzyme A on Serum Lipids in Patients With Hyperlipidemia: a Randomized, Double-blinded, Placebo-controlled, Multi-center Clinical Trial
Brief Title: The Effects of Coenzyme A on Serum Lipids in Patients With Hyperlipidemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Jiangtao Lai, MD, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008MMXX2CoA005
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Hyperlipoproteinemia
MeSH Terms: conditions — Hyperlipoproteinemias | interventions — Coenzyme A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Coenzyme A 200mg (Active Comparator): Coenzyme A 200mg per day.
  Interventions: Drug: Coenzyme A
- Placebo (Placebo Comparator): Capsule without coenzyme A.
  Interventions: Drug: Placebo
- Coenzyme A 400mg (Active Comparator): Coenzyme A 400mg per day.
  Interventions: Drug: Coenzyme A

INTERVENTIONS:
Drug: Coenzyme A — Coenzyme A 200mg per day.
  Other Names: Low dose coenzyme A therapy.
  Arms: Coenzyme A 200mg
Drug: Coenzyme A — Coenzyme A 400mg per day.
  Other Names: High dose coenzyme A therapy.
  Arms: Coenzyme A 400mg
Drug: Placebo — Capsule without coenzyme A.
  Other Names: Controls.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the lipid lowering effects and clinical safety of a natural hypolipidemic compound, coenzyme A （CoA） capsule in Chinese patients with moderate dyslipidemia.

DETAILED DESCRIPTION:
Hyperlipidemia plays important roles in the development and progression of atherosclerosis. Modulating lipid levels has been shown to reduce the development of atherosclerosis and incidence of cardiovascular disease. The HMG-CoA reductase inhibitors (also known as statins) are the most effective agents available in the management of hyperlipidemia and prevention of major cardiovascular events. Although statin based therapy is commonplace in primary and secondary prevention, several economical, clinical and safety issues have been raised, so that there is ongoing research into new, safer and more effective agents to be used alone or in combination with existing cardiovascular drugs.

Coenzyme A (CoA) is a ubiquitous essential cofactor that plays a central role in the metabolism of carboxylic acids, including short- and long-chain fatty acids, as well as carbohydrate and protein. In the metabolic pathway of lipid, CoA participates in fatty acid β-oxidation, promoting triglyceride (TG) catabolism. Previous research revealed that insufficiency of CoA in vivo influenced fatty acid β-oxidation catabolism and impaired clearance of TG from plasma, which was supposed to be one plausible reason resulting in type Ⅱb and Ⅳ hyperlipoproteinemia. In addition, epidemiological studies showed the prevalence of serum lipids level increased with age, which may be related to the reduction of CoA synthesis in aging individuals. Moreover, studies on animals have given evidence to prove that supplement of CoA had normalizing activity on plasma lipids in dyslipidemia.

Pantethine is a versatile and very well tolerated hypolipidemic agent that can decrease serum triglycerides, LDL cholesterol, and apolipoprotein B, while increasing HDL cholesterol and apolipoprotein A-I. Pantethine is the disulfide of pantetheine which per se occurs naturally as a product of coenzyme A catabolism. Theoretically, antihyperlipidemia effect of CoA should be more directly and effectively than pantethine. Researches on rabbits and rats models prove that high dose CoA orally can relieve fasting hyperlipidemia and insulin resistance induced by high fat diet. So far there has not been sufficient clinical research data to support the efficacy of CoA in dyslipidemia patients. The present study shows, for the first time, the safety, effectiveness of oral CoA.

ELIGIBILITY:
Inclusion Criteria:

* TG 2.3～6.5mmol/l meeting the China National Cholesterol Education Programme diagnostic criteria of hyperlipidemia.

Exclusion Criteria:

1. TC >7.5 mmol/l or LDL-C >3.6 mmol/l
2. Body Mass Index > 30 kg/m2
3. drug induced secondary hypercholesterolemia (such as dibenzothiazine, contraceptive agent or adrenal cortex hormone)
4. pregnancy
5. acute coronary syndrome, acute myocardial infarction or undergone a revascularization procedure within 6 months
6. acute liver disease or hepatic dysfunction, as determined by levels of alanine aminotransferase (ALT) or aspartate aminotransferase levels (AST) more than 3-fold the upper normal limit
7. nephrotic syndrome or serum creatinine (Cr) (≥179 µmol/L) and creatine phosphokinase (CK) more than 3-fold the upper normal limit
8. primary hypothyroidism
9. psychiatric patients and HIV-infected patients
10. poorly controlled hypertension, as indicated by a Systolic Blood Pressure >180 mmHg or Diastolic Blood Pressure >110 mmHg
11. Type I diabetes mellitus（DM）, poorly controlled Type II DM (BS>11.0 mmol/L ) or Type II DM with LDL-C >2.6 mmol/L.Patients using immunosuppressive drugs, prohibited medication or other lipid-lowing drugs were also excluded. Subjects were also ineligible for the study if they had any severe disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The changes of TG levels. | 4 and 8 weeks after administration.

SECONDARY OUTCOMES:
The changes of TC, LDL-C, and HDL-C levels. | 4 and 8 weeks after administration.

CONTACTS AND LOCATIONS:
Overall Officials: Junzhu Chen, MD, Principal Investigator — Zhejiang University